CLINICAL TRIAL: NCT07249177
Title: Validity and Reliability of the Upper Extremity Functional Index in Patients With Carpal Tunnel Syndrome
Brief Title: Upper Extremity Functional Index in Carpal Tunnel Syndrome
Status: Completed | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, UMUT ERASLAN, Assistant Professor, Pamukkale University
Other Study IDs: E-60116787-020-28687
Record Dates: First submitted 2025-11-17; First posted 2025-11-25 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Carpal Tunnel Syndrome (CTS); Upper Extremity Function
Keywords: psychometrics; carpal tunnel syndrome; outcome measures; upper extremity functional index
MeSH Terms: conditions — Carpal Tunnel Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients aged 18-65 years diagnosed with carpal tunnel syndrome.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — The Upper Extremity Functional Index (at the first session and after 2 weeks), the Michigan Hand Outcomes Questionnaire and the Boston Carpal Tunnel Questionnaire were administered to patients using a face-to-face assessment method.

SUMMARY:
The aim of this study was to investigate the validity and reliability of the Upper Extremity Functional Index in patients with carpal tunnel syndrome. This cross-sectional study included 101 patients diagnosed with carpal tunnel syndrome at a university hospital. Patients were administered the Upper Extremity Functional Index, Michigan Hand Outcomes Questionnaire, and Boston Carpal Tunnel Questionnaire surveys. Test-retest reliability, internal consistency, and construct validity of the Upper Extremity Fuctional Index were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* To be diagnosed with carpal tunnel syndrome, to be a volunteer, and to be between the ages of 18 and 65 years.

Exclusion Criteria:

* no history of other trauma, disease or surgery in the affected limb and difficulty communicating

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study included patients aged 18-65 years who were diagnosed with carpal tunnel syndrome after visiting the neurology outpatient clinic of a university hospital, who volunteered, who had no history of other trauma, disease, or surgery in the affected limb, and who had no communication difficulties. The patients were included before starting any conservative or surgical treatment programme.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2021-06-28 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2022-11-18 (Actual)

PRIMARY OUTCOMES:
Upper Extremity Functional Index | The questionnaire was administered at baseline (after diagnosis of carpal tunnel syndrome) and 15 days after the baseline assessment.
  It is a 20-item scale scored using a 4-point Likert scale (0 = Extremely difficult/I cannot do it, 4 = I do not experience any difficulty). The patient scores between 0 and 80, and it is recommended that the total score be used in studies. A high score indicates that the patient has good upper extremity function.
Michigan Hand Outcomes Questionnaire | The questionnaire was administered at baseline (after diagnosis of carpal tunnel syndrome)
  This questionnaire evaluates the functionality of the hand and consists of 63 questions in total. Each question is scored between 1-5 and the score of each section varies between 0-100. High total score indicates high satisfaction.
Boston Carpal Tunnel Questionnaire | The questionnaire was administered at baseline (after diagnosis of carpal tunnel syndrome)
  It has been developed to assess the severity of symptoms and functional status in patients with carpal tunnel syndrome. The symptom severity scale consists of 11 questions, while the functional status scale consists of 8 questions. Each question is scored between 1 and 5. A higher symptom severity or functional status score indicates worse symptoms or functional impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aytar A, Yuruk ZO, Tuzun EH, Baltaci G, Karatas M, Eker L. The Upper Extremity Functional Index (UEFI): cross-cultural adaptation, reliability, and validity of the Turkish version. J Back Musculoskelet Rehabil. 2015;28(3):489-95. doi: 10.3233/BMR-140545. PMID 25322741
- [Background] Sousa RL, Moraes VY, Zobiole AF, Nakachima LR, Belloti JC. Diagnostic criteria and outcome measures in randomized clinical trials on carpal tunnel syndrome: a systematic review. Sao Paulo Med J. 2023 Apr 17;141(6):e2022086. doi: 10.1590/1516-3180.2022.0086.07022023. eCollection 2023. PMID 37075455